CLINICAL TRIAL: NCT01775384
Title: Influence of a Polyphenol-enriched Protein Powder on Exercise-induced Inflammation and Oxidative Stress in Athletes: a Metabolomics Approach
Brief Title: Polyphenols, Exercise, and Metabolomics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Appalachian State University (Other)
Collaborators: Dole Food Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12-0134
Record Dates: First submitted 2013-01-02; First posted 2013-01-25 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Exercise-induced Inflammation; Exercise-induced Oxidative Stress; Exercise-induced Immune Dysfunction
Keywords: Inflammation; Oxidative stress; Immune dysfunction; Metabolomics.
MeSH Terms: conditions — Inflammation; Immune System Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nutrasorb (Experimental): Soy protein powder sorbed with polyphenols from blueberries and green tea extract
  Interventions: Dietary Supplement: Nutrasorb
- Placebo (Placebo Comparator): Soy protein isolate powder without polyphenols (with food coloring)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Nutrasorb — from blueberry and green tea extracts (2,136 mg/d gallic acid equivalents)
  Arms: Nutrasorb
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Nutrasorb is a newly developed food product (see www.nutrasorb.com). This study will use the Nutrasorb soy protein product that is matrixed with polyphenols from blueberries and green tea extract, and test for efficacy as a nutritional countermeasure to exercise-induced physiologic stress (i.e., immune dysfunction, inflammation, and oxidative stress) using both traditional and metabolomics-based outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Male or female endurance athletes; competitive runners or cyclists
* Capable of exercising for 2.5 h at a high intensity in the lab
* Ages 18-55
* Agree to train normally and stay weight stable.
* Agree to avoid the use of large dose vitamin/mineral supplements
* Agree to avoid herbs and medications that influence inflammation

Exclusion Criteria:

* Regularly take supplements or medicines known to effect inflammation.
* At moderate or high risk for cardiovascular disease.
* Younger than 18 or older than 55 years of age.
* No history of competing in long distance running and cycling races.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2012-04; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Metabolomics; change in metabolites over time | 18-day period; Blood samples collected pre- and post-14 d supplementation, and immediately and 14 h after the third day of running
  GC-MS and LC-MS through Metabolon

SECONDARY OUTCOMES:
Change in inflammation | 18-day period; Blood samples collected pre- and post-14 d supplementation, and immediately and 14 h after the third day of running
  CRP and a cytokine panel
Change in oxidative stress | 18-day period; Blood samples collected pre- and post-14 d supplementation, and immediately and 14 h after the third day of running
  F2-isoprostanes, protein carbonyls, FRAP, ORAC
Change in immune function | 18-day period; Blood samples collected pre- and post-14 d supplementation, and immediately and 14 h after the third day of running
  Anti-viral activity using virus-infected HeLa cells

CONTACTS AND LOCATIONS:
Overall Officials: David C Nieman, DrPH, Principal Investigator — Appalachian State University
Locations (1):
- ASU Human Performance Laboratory, North Carolina Research Campus, Kannapolis, North Carolina, United States

REFERENCES:
- [Derived] Nieman DC, Gillitt ND, Knab AM, Shanely RA, Pappan KL, Jin F, Lila MA. Influence of a polyphenol-enriched protein powder on exercise-induced inflammation and oxidative stress in athletes: a randomized trial using a metabolomics approach. PLoS One. 2013 Aug 15;8(8):e72215. doi: 10.1371/journal.pone.0072215. eCollection 2013. PMID 23967286
- See also: Lab web site — http://www.ncrc.appstate.edu